CLINICAL TRIAL: NCT02222051
Title: Tai Chi for Chronic Non-specific Neck Pain: A Randomized Controlled Trial
Brief Title: Tai Chi for Chronic Non-specific Neck Pain
Acronym: TaiChiNe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, PhD, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-5672 Tai Chi Neck Pain
Record Dates: First submitted 2014-08-18; First posted 2014-08-21 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Neck Pain
Keywords: neck pain; chronic pain
MeSH Terms: conditions — Neck Pain; Chronic Pain | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tai Chi (Experimental): Simplified 24 Yang Style 12 weeks, 1x/week, 60-90 minutes
  Interventions: Behavioral: Tai Chi
- Neck exercise (Active Comparator): conventional neck exercises 12 weeks, 1x/week, 60 min stretching and strengthening, neck education
  Interventions: Behavioral: Neck exercises
- Usual care (No Intervention): Usual care, no specific study intervention this group is offered Tai Chi or neck exercises at the end of the study

INTERVENTIONS:
Behavioral: Tai Chi — traditional chinese martial art meditative movement technique
  Other Names: Taiji; T'ai Chi
  Arms: Tai Chi
Behavioral: Neck exercises — group exercises for strengthening and stretching neck and back muslces to alleviate neck pain
  Other Names: neck training
  Arms: Neck exercise

SUMMARY:
In this study the efficacy of Tai Chi will be tested in comparison to conventional neck exercises and usual care in a randomized controlled trial. Tai Chi and neck exercises will be lead by a trained exercise therapist and Tai Chi instructor, both groups receive 12 weeks of training, once weekly for 60-90 min in a group setting. Pain, Disability, quality of life, wellbeing, stress perception, psychological distress will be used to determine effects.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* chronic non specific neck pain (3 months at least)
* 45mm pain intensity on average on the visual analog scale

Exclusion Criteria:

* specific neck pain due to
* inflammatory diseases
* rheumatic diseases
* neurological diseases
* prolapse or protrusion
* oncological disease
* trauma (whiplash)
* congenital deformity of the spine
* severe comorbidity (somatic, psychiatric)
* pregnancy
* participation in other clinical trials
* regular practice of tai chi, qigong, yoga in the past 6 months
* medication with opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
pain intensity | week 12
  pain intensity on a visual analogue scale (0-100mm)

SECONDARY OUTCOMES:
pain intensity | week 24
  pain intensity on a visual analogue scale (0-100mm)
pain on movement | week 12, week 24
  pain intensity on a visual analogue scale (0-100mm) evoked by head movement into 6 directions POM validated by Lauche et al., 2014, Pain Medicine
neck disability | week 12, week 24
  neck disability index (NDI), Vernon et al.
health related quality of life | week 12, week 24
  short form quality of life questionnaire (SF-36), Bullinger and Kirchberger
Anxiety and Depression | week 12, week 24
  Hospital Anxiety and Depression Scale (HADS)
Wellbeing | week 12, week 24
  Wellbeing on the FEW16 Questionnaire
Stress | week 12, week 24
  Subjective stress perception, Perceived Stress Scale (PSS)
interoceptive awareness | week 12, week 24
  The Multidimensional Assessment of Interoceptive Awareness (MAIA)
Postural Awareness | week 12, week 24
  Postural Awareness Questionnaire (PAS)
Safety | week 24
  All adverse and serious adverse events
pain intensity ratings | week 12
  daily rating of pain intensity, visual analog scales
use of analgetics | week 12
  daily information on use of analgetics
use of concomitant therapies | week 12
  daily information on use of concomitant therapies for neck pain

OTHER OUTCOMES:
Experiences | Week 24
  Experiences with Tai Chi and neck exercises, qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof., Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Lauche R, Wayne PM, Fehr J, Stumpe C, Dobos G, Cramer H. Does Postural Awareness Contribute to Exercise-Induced Improvements in Neck Pain Intensity? A Secondary Analysis of a Randomized Controlled Trial Evaluating Tai Chi and Neck Exercises. Spine (Phila Pa 1976). 2017 Aug 15;42(16):1195-1200. doi: 10.1097/BRS.0000000000002078. PMID 28146026
- [Result] Lauche R, Stumpe C, Fehr J, Cramer H, Cheng YW, Wayne PM, Rampp T, Langhorst J, Dobos G. The Effects of Tai Chi and Neck Exercises in the Treatment of Chronic Nonspecific Neck Pain: A Randomized Controlled Trial. J Pain. 2016 Sep;17(9):1013-27. doi: 10.1016/j.jpain.2016.06.004. Epub 2016 Jun 23. PMID 27345663
- [Derived] Allende S, Cramer H, Wayne P, Lauche R. Investigating Inter- and Intra-individual Differences in Tai Chi Practice Time, Pain, and Mood Among Participants with Chronic Nonspecific Neck Pain: Secondary Analysis of a Randomized Controlled Trial. J Integr Complement Med. 2023 Apr;29(4):234-240. doi: 10.1089/jicm.2022.0789. Epub 2023 Mar 17. PMID 36930781